CLINICAL TRIAL: NCT06745856
Title: A Trial of Intraoperative 5-fluorouracil in Primary Glaucoma Filtration Surgery: Effects on Long Term Intraocular Pressure Control and Disease Progression
Brief Title: Intraoperative 5-fluorouracil Augmentation of Trabeculectomy
Acronym: MoreFlow
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Moorfields Eye Hospital NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: G9330070
Record Dates: First submitted 2023-12-22; First posted 2024-12-20 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Glaucoma; Primary Open Angle Glaucoma
Keywords: glaucoma; trabeculectomy; intraocular pressure; randomized control study; antimetabolite; 5 fluorouracil
MeSH Terms: conditions — Glaucoma; Glaucoma, Open-Angle | interventions — Fluorouracil; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 5-fluorouracil (Active Comparator): antimetabolite to prevent wound healing
  Interventions: Drug: 5-fluorouracil
- placebo (Placebo Comparator): Subconjunctival placebo.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: 5-fluorouracil — Subconjunctival, peroperative, application of 50mg/ml concentration of 5-fluoruracil.
  Other Names: 5 fluorouracil subconjunctival injection
  Arms: 5-fluorouracil
Drug: placebo — Subconjunctival, peroperative application of normal saline (NaCl 0.9%)
  Other Names: sodium chloride solution (0.9%)"
  Arms: placebo

SUMMARY:
5-fluorouracil (5FU) is an antimetabolite that has been demonstrated to have beneficial effects when injected into the subconjunctival space after glaucoma surgery (trabeculectomy). The hypothesis of this study is that a similar beneficial effect can be achieved with a single intraoperative application of 5FU. This hypothesis is tested with a randomized control study.

DETAILED DESCRIPTION:
Glaucoma is the commonest cause of irreversible blindness worldwide. Treatment is initially with topical medication, but when the intraocular pressure is still poorly controlled, surgical treatment is required. The surgical treatment of choice remains the trabeculectomy and this is often augmented with antimetabolite.

The choice of antimetabolite varies between surgeons, as does the indications for use. Postoperative delivery of the drug can be uncomfortable for the patient and time consuming. This study examines the potential benefits and side effect profile of intraoperative 5FU compared to unaugmented trabeculectomy.

The patients are recruited from Moorfields Eye Hospital and followed up by the staff from the glaucoma department.

ELIGIBILITY:
Inclusion Criteria:

* A measured intraocular pressure > or equal to 22 mm Hg on at least one visit before the time of listing for surgery and while on the current drop regime.
* The ability to complete a Humphrey 24-2 visual field test with <20% false positives, <33% false negatives and <20% fixation losses, and the presence of 2 locations > 5decibels (dB) less than normal or one location >10 dB less than normal.
* The presence of a focal or diffuse area of optic disc rim loss, as shown by a reduction of optic rim thickness to less than one tenth of disc diameter at any point on the disc. (alternatively, optic disc which in the opinion of the patient's consultant shows glaucomatous changes as shown by focal or diffuse optic rim thinning)

Exclusion Criteria:

* Anterior segment neovascularisation
* Any intraocular epithelial ingrowth
* Retinal or optic nerve neovascularisation
* Aphakia
* Previous glaucoma filtering surgery
* Uveitis
* Any previous intraocular surgery
* Inability or unwillingness to give informed consent
* Inability or unwillingness to return for postoperative follow-up as prescribed in the trial regimen
* Unwillingness to accept randomisation
* Patient less than 40 years of age
* Chemotherapy in the 6 weeks prior to surgery
* Any other disease causing visual field loss or likely to cause field loss over the next three years e.g. diabetic retinopathy, pituitary disease or stroke.
* Pregnancy or female of childbearing age who may be pregnant at time of treatment. A pregnancy test will be performed on all women of childbearing age to rule out pregnancy.
* Cataract that is deemed significant enough to require surgery during the course of the trial or that makes field testing or optic disc recording by either photography or the scanning laser ophthalmoscope unreliable or not technically possible.
* Any medical condition likely to prevent the patient from regularly attending for the next three years
* Previous conjunctival surgery at proposed site of trabeculectomy
* Chronic use of topical or systemic steroids
* Previous squint surgery

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 368 (Actual)
Dates: Start 1996-04; Primary Completion 2000-06 (Actual); Study Completion 2003-06 (Actual)

PRIMARY OUTCOMES:
Glaucoma control | a minimum of 3 years follow up
  Raised Intra Ocular Pressure (IOP) of >21 millimetres of mercury (mmHg) on two or more consecutive visits recorded at the end of a visit following any physical intervention. Visual field progression that met a modified criteria of the Collaborative Normal Tension Glaucoma Study (CNTGS). Optic disc cupping progression identified by the examining clinician and confirmed with stereo-photographic documentation of the optic nerve neuroretinal rim changes read by two masked examiners. If any of these outcome measures were reached, the patient was classified as a 'trial failure' and then treated further depending on the clinicians discretion.

SECONDARY OUTCOMES:
long term safety of intraoperative 5FU | a minimum of 3 years follow up
  A secondary objective was to examine the relationship between IOP control and glaucoma progression. IOP failure was defined in four categories ≤ 14mmHg, ≤ 17mmHg, ≤ 21mmHg or > 21mmHg. It was hypothesized that when compared to placebo, intraoperative 5FU would result in lower IOP levels and better control of IOP for at least 3 years reducing the risk of progression of visual field loss or optic nerve damage.